CLINICAL TRIAL: NCT06408428
Title: Glioma Intraoperative MicroElectroCorticoGraphy
Acronym: MicroECoGG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: PANAXIUM (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: C20-90
Record Dates: First submitted 2024-01-23; First posted 2024-05-10 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Glioma; Epilepsy
Keywords: Glioma surgery; Awake surgery; MicroElectroCorticoGraphy; EEG
MeSH Terms: conditions — Glioma; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Glioma Surgery - MicroECoG recording (Experimental)
  Interventions: Device: PANAXIUM MicroECoG

INTERVENTIONS:
Device: PANAXIUM MicroECoG — The PANAXIUM microelectrode ( 4x2 cm, 6 micron-thick electrode comprising 128 electrodes (28 500 µm electrodes, 96 30 µm diameter microelectrodes organized as tetrodes and 4 reference electrodes) will be placed on the cortical surface and repositioned every 90 seconds to sample the entire exposed brain surface. During the cortical electrical stimulation mapping phase, the electrode will be left at the edge of the field to detect epileptic discharges induced by stimulation. After resection, a new recording of the residual cortical surface will be made to check for persistent electrical anomalies. In the last 10 patients, the Panaxium microECoG will be compared with a macro-electrode for clinical use.

SUMMARY:
The goal of this clinical trial is to validate the safety and to assess the quality of the signals provided by newly developed micro ElectroCorticoGraphy electrodes, provided by the company Panaxium, based on conductive polymers (PEDOT:PSS) in patients suffering of gliomas during resection surgery performed in awake condition. The main questions it aims to answer are:

* Safety of PEDOT:PSS microECoGs by assessing the rate of serious adverse events associated with their use during glioma surgery.
* Quality of PEDOT:PSS microECoGs recordings, as compared with recordings with traditional macroelectrodes, assessed by signal-to-noise ratio, impedance, ability to detect ripples (100-250 Hz) and fast ripples (250-600 Hz), ability to record epileptic activity (spikes and equivalent) either spontaneously or following direct electrical stimulation (afterdischarges).
* Practicality of microelectrodes use as perceived by neurosurgeons.
* Exploratory objectives: ability to record multi-unit activity, correlation between microECoG activity and tumor infiltration - local oncometabolite concentrations, determination of epileptic seizure rate during electrode use.

Participants will be recorded during awake glioma surgery by the newly developed micro ElectroCorticoGraphy electrodes and by routine macroelectrodes, as standard of care during both mapping of cortical activities and electrical stimulations used to assess the functional mapping mandatory for tailored tumor resection.

DETAILED DESCRIPTION:
Electroencephalography (EEG) is a widely-used tool for studying brain activity, developed in humans in the late 1920s. Its indications have evolved as brain imaging techniques have developed, but it remains extremely useful in the fields of epileptology, comas, brain death, post-anoxic, metabolic, toxic encephalopathies and encephalitis. Alongside scalp EEG, intracranial recordings have been developed to optimize the localization of epileptic activity, with a view to epilepsy surgery.

Two main categories of intracranial electrodes are currently in use.

1. StereoElectroEncephalopGraphy electrodes consist of a stylus with a string of cylindrical contacts along its length, implanted directly into the brain parenchyma.
2. ElectroCorticoGraphy (ECoG) electrodes, non-penetrating, organized in strips or grids of 4 to 64 electrodes, disc-shaped, 0.2 to 1 cm in diameter, 0.5 to 1 mm thick, used to collect cerebral activity at the cortical surface.

Among its indication, surgery is a favorable circumstance for using ECoG. During brain surgery, cortical exposure enables cortical EEG recording without additional invasiveness. Intraoperative ECoG is of particular interest in epilepsy surgery, recently reactivated by the discovery of better electrophysiological biomarkers. In glioma surgery, often performed under awake conditions, cortical recording helps to establish a functional cerebral map and to adapt the resection. Indeed, ECoG recordings can be performed during awake surgery, without any disturbance of neuronal activity by anesthesia, to map epileptic activity (using visual identification of spikes) and to look for seizures induced by electrical stimulation. The evolution of these recording techniques is moving towards the development of tools for automatic analysis and mapping of new biomarkers, more relevant but more difficult to record because they are more focal and characterized by amplitudes close to background noise, such as high-frequency oscillations. New types of cortical electrodes are being developed to improve the spatial resolution (better localization), temporal resolution (faster activity detection) and detection sensitivity (signal-to-noise ratio) of cortical electrical signals.

New electrodes have recently been developed, based on the use of conductive organic polymer coatings such as poly(3,4-ethylenedioxythiophene (PEDOT: PSS), to optimize the signal-to-noise ratio, organized in electrode arrays that are 100 times thinner (5 microns vs. 0.5 mm for standard electrodes), 250 times smaller (between 30 and 500 microns vs. 8 mm for standard electrodes) and with more electrodes (128 vs. 6 or 8 for standard electrodes). This type of electrode, known as microECoG, has been validated in animals and has already been used in human research for intraoperative cortical recordings. They enable us to improve the quality of the recorded signal and to go down to a new scale, at the level of the neuron. Moreover, the very low thickness of the electrodes improves their conformability to the cortex, making them much more tolerable and enabling extended recordings to be envisaged as part of future man/machine interfaces.

The French company Panaxium is developing microECoG electrodes. As part of a collaborative project, Panaxium have designed a 4x2 cm, 6 micron-thick electrode comprising 128 electrodes (28 500 µm electrodes, 96 30 µm diameter microelectrodes organized as tetrodes and 4 reference electrodes) for clinical use in humans. The aim of this study is to explore the safety and quality of signals collected by the Panaxium microECoG during awake surgery for brain gliomas. Recording will be carried out using a high-performance EEG system CE-marked for medical use in humans.

The electrode will be placed on the cortical surface and repositioned every 90 seconds to sample the entire exposed brain surface. During the cortical electrical stimulation mapping phase, the electrode will be left at the edge of the field to detect epileptic discharges induced by stimulation. After resection, a new recording of the residual cortical surface will be made to check for persistent electrical anomalies. The surgeries and recordings will be carried out in 3 centers by neurosurgeons with expertise in brain tumors and awake surgery: Hôpital Sainte-Anne/GHU Paris), Hôpital Pietié-Salpêtrière, Hopital Fondation Adolphe de Rostschild. In the last 10 patients, the Panaxium microECoG will be compared with a macro-electrode for clinical use.

The primary endpoint will be the incidence of Serious Adverse Events due to the use of Panaxium microelectrodes during surgery and the following four days: cortical lesion by the electrode, infection, bleeding, aseptic meningitis, neurological deficit due to the use of the electrode, death. Secondary evaluation criteria will be the quality of recordings enabled by the Panaxium microECoG (signal-to-noise ratio reflecting signal quality, electrode impedance during surgery reflecting technical quality, detection of fast ripple (100-250 Hz) and fast ripple (250-600 Hz) oscillations), only possible with high-performance recorders, ability to record spontaneous epileptic activity (spikes and equivalent) or direct post-electrical stimulation (post-discharges)) and practicality of use as perceived by neurosurgeons. Finally, as an exploratory study for future uses of these electrodes, we will investigate their ability to record multi-unit activity (action potentials from single neurons) and the correlation between recorded activity and tumor infiltration, as well as local oncometabolite concentration.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering of a diffuse cerebral glioma for which surgical resection is indicated.
* Planned awake surgery with intraoperative functional mapping.
* Planned surgery with ECoG electrophysiological monitoring.
* Age greater than or equal to 18 years.
* Enrolled in a social security scheme, Couverture Médicale Universelle (CMU) or equivalent.
* Have given written consent.

Exclusion Criteria:

* Acute or untreated infection (viral, bacterial or fungal).
* Current treatment with antibiotics.
* Pregnant or breast-feeding women.
* Other pathologies that could interfere with the neurological evaluation or compromise the subject's safety.
* Participation in therapeutic biomedical research that could modify the lesion or its environment during the study period (whether by drug or medical device) or subject to an exclusion period for other research.
* Adult subject to legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Safety of PEDOT:PSS microECoGs use | 30 months
  Assessment of the safety of PEDOT:PSS microECoGs use by assessing the rate of serious adverse events associated with their use during glioma surgery

SECONDARY OUTCOMES:
Quality of PEDOT:PSS microECoGs recordings | 30 months
  Quality of PEDOT:PSS microECoGs recordings assessment by signal-to-noise ratio, impedance, ability to detect ripples (100-250 Hz) and fast ripples (250-600 Hz), ability to record epileptic activity (spikes and equivalent) either spontaneously or following direct electrical stimulation (afterdischarges)
Practicality of microelectrodes use as perceived by neurosurgeons. | 30 months
  Practicality of microelectrodes use as perceived by neurosurgeons.

OTHER OUTCOMES:
ability to record multi-unit activity, correlation between microECoG activity and tumor infiltration - local oncometabolite concentrations, determination of epileptic seizure rate during electrode use | 30 months
  ability to record multi-unit activity, correlation between microECoG activity and tumor infiltration - local oncometabolite concentrations, determination of epileptic seizure rate during electrode use

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Huberfeld, MD, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (3):
- France (3):
  - Hôpital Pitié Salpêtrière, Paris
  - Centre Hospitalier Sainte-Anne, Paris
  - Hôpital Fondation Adolphe de Rothschild, Paris

IPD SHARING:
Plan to Share IPD: No